CLINICAL TRIAL: NCT01278095
Title: A Randomized, Open Label, 3-way Crossover Study to Compare the Oral Bioavailability of GLPG0555 After Single-dose Intake in Healthy Subjects as a Solid Dispersion Formulation, With and Without Food, Relative to a Nanosuspension Formulation
Brief Title: Oral Bioavailability of GLPG0555 in Different Solid Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Senior Vice President Development, Galapagos
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: GLPG0555-CL-103; 2010-022457-42 (EudraCT Number)
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2011-03

CONDITIONS: Healthy
Keywords: Safety; Tolerability; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- GLPG0555 solid dispersion, fasting (Experimental): 50 mg as solid dispersion capsule, in fasting condition
  Interventions: Drug: GLPG0555 solid dispersion
- GLPG0555 solid dispersion, fed (Experimental): 50 mg as solid dispersion capsule, after breakfast
  Interventions: Drug: GLPG0555 solid dispersion
- GLPG0555 nanosuspension, fed (Experimental): 50 mg as nanosuspension, given after breakfast
  Interventions: Drug: GLPG0555 nanosuspension

INTERVENTIONS:
Drug: GLPG0555 solid dispersion — solid dispersion capsules, 50 mg, single dose
  Arms: GLPG0555 solid dispersion, fasting; GLPG0555 solid dispersion, fed
Drug: GLPG0555 nanosuspension — Nanosuspension, 50 mg, single dose
  Arms: GLPG0555 nanosuspension, fed

SUMMARY:
The purpose of the study is to compare the pharmacokinetics of a solid capsule formulation of GLPG0555 with a nanosuspension, and to assess safety and tolerability of a single dose of GLPG0555.

ELIGIBILITY:
Inclusion Criteria:

* healthy male
* BMI between 18-30 kg/m², inclusive.

Exclusion Criteria:

* significantly abnormal platelet function or coagulopathy
* smoking
* drug or alcohol abuse

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-01; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Bioavailability of solid formulation | 72 hrs

SECONDARY OUTCOMES:
Safety and tolerability of single doses of GLPG0555 | up to 10 days postdose

CONTACTS AND LOCATIONS:
Overall Officials: Gerben van 't Klooster, PhD, Study Director — Galapagos NV; Jos Leempoels, MD, Principal Investigator — SGS Stuivenberg
Locations (1):
- SGS Stuivenberg, Antwerp, Belgium